CLINICAL TRIAL: NCT06481631
Title: Empowering Women for Postpartum Care and Reproductive Health in Mississippi Delta
Brief Title: Patient-clinical Linkages to Improve Trust and Engagement in Postpartum Healthcare
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jackson State University (Other)
Collaborators: Mississippi State Department of Health (Other Government); University of Mississippi Medical Center (Other); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1U54HD113238-02 (NIH)
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-06

CONDITIONS: Family Dynamics; Trust in Healthcare System; Family Structure; Health Literacy; Contraception; Maternal Behavior; Postpartum Mood Disturbance

STUDY DESIGN:
Intervention Model Description: Clinical trial with one arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PEN-3 Assessment Model (Other): Application of a sociocultural model to assess patient-clinical linkages that support positive maternal health outcomes
  Interventions: Behavioral: The PEN-3 Intervention Model

INTERVENTIONS:
Behavioral: The PEN-3 Intervention Model — The PEN-3 Model is a sociocultural model for planning and assessing participant behavior within the context a cultural phenomenon. It will be used to assess intervention impact on patient-clinical linkages in the Mississippi Delta.

SUMMARY:
Maternal mortality in the United States is higher than in peer nations and has not decreased since 1990. Beyond mortality, severe maternal mortality impacts far too many women. Not only are these high rates alarming, but notable racial/ethnic and socioeconomic disparities exist. These inequities are highly regional, with women living in the rural southeast part of the United States, including the Mississippi Delta, having the highest rates of maternal mortality and morbidity. Unfortunately, these disparities have proven to be stubbornly resistant to interventions, necessitating an innovative multifaceted approach focused on community practice, building trust, and prioritizing patient voices. To meet this need, this proposal aims to establish the Mississippi Delta Research Center of Excellence for Maternal Health with the goal of addressing preventable maternal mortality, decreasing severe maternal morbidity, and promoting maternal health equity in partnership with the Mississippi Delta community. This patient-clinical linkages intervention study will evaluate the effectiveness of a multilevel and multisector communication and health literacy strategy to increase trust and engagement in postpartum healthcare among women in the Mississippi Delta, with a specific focus on Black women, their families, and their communities.

These research projects both have the overarching goal of partnering with the community to determine and meet the needs of pregnant and postpartum women in the Mississippi Delta and address the disparities within maternity health and health care outcomes.

DETAILED DESCRIPTION:
Maternal mortality in the United States is higher than in peer nations and has not decreased since 1990. Beyond mortality, severe maternal mortality impacts far too many women. Not only are these high rates alarming, but notable racial/ethnic and socioeconomic disparities exist. These inequities are highly regional, with women living in the rural southeast part of the United States, including the Mississippi Delta, having the highest rates of maternal mortality and morbidity. Unfortunately, these disparities have proven to be stubbornly resistant to interventions, necessitating an innovative multifaceted approach focused on community practice, building trust, and prioritizing patient voices. To meet this need, this proposal aims to establish the Mississippi Delta Research Center of Excellence for Maternal Health with the goal of addressing preventable maternal mortality, decreasing severe maternal morbidity, and promoting maternal health equity in partnership with the Mississippi Delta community. This research center will conduct two multi-layered research projects. Research Project 1 will determine the effectiveness of an evidenced-based community health worker home visiting program grounded in extensive patient and community participation. Research Project 2 will evaluate the effectiveness of a multilevel and multisector communication and health literacy strategy to increase trust and engagement in postpartum healthcare among women in the Mississippi Delta, with a specific focus on Black women, their families, and their communities. These research projects both have the overarching goal of partnering with the community to determine and meet the needs of pregnant and postpartum women in the Mississippi Delta and address the disparities within maternity care.

ELIGIBILITY:
Inclusion Criteria:

* Identified as high risk pregnancy
* Postpartum mothers/parents 18-45 years
* Resident of the one of 5 target counties (Washington, Bolivar, Scott, Humphreys, and Carroll)
* Maternal healthcare providers in target counties
* Maternal community health leaders

Exclusion Criteria:

* not identified as high risk pregnancy
* 18 years of age postpartum
* cesarean birth
* non-resident of the 5 target counties

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — biological women at birth; women who have vaginal deliveries
Enrollment: 250 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Improve trust in the healthcare system | 12 months from consent to participate
  Mixed methods approach using Trust in Physician Scale & Researcher developed qualitative tool
Increase maternal health literacy (patient and provider perspectives) | 12 months from consent to participate in the intervention
  Brief literacy screening tool to evaluate health literacy in the health system (Qualitative and Quantitative Measures
Increase engagement in the maternal health care system (patient-clinic linkages) | 12 month from consent to participation in the intervention
  Contraceptive Counseling measure tool to evaluate the patient experiences with provider care and vice-versa; minimally 2 post-partum clinec visits in postpartum period
Strengthen structuring of family support systems | 12 months from consent to participation in the intervention
  Family crisis coping response (F-COPES) measure to determine patient (mother) and family perceptions and experiences with structuring family support fo postpartum care period.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Shaw, PhD, Principal Investigator — Jackson State University; Mary Shaw, PHD, M.ED, Study Director — Jackson State University
Locations (1):
- Jackson State University/Department of Behavioral & Environmental Health, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No